CLINICAL TRIAL: NCT01347359
Title: Peer to Peer Mentoring For Individuals With Early Inflammatory Arthritis: An Effectiveness Study (Pilot RCT)- Peer Mentoring Program
Acronym: P2P EIA RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Rheumatology Association (Other); Mount Sinai Hospital, Canada (Other); The Arthritis Society, Canada (Other); Unity Health Toronto (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Dr. Mary Bell, Rheumatologist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 094-2011
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Early Inflammatory Arthritis
Keywords: Peer support; Peer mentoring; Peer counselling; Arthritis; Inflammatory arthritis; Early inflammatory arthritis; Rheumatoid arthritis; Chronic disease
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid; Chronic Disease | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- One-on-one peer support (Experimental): The peer support intervention will take the form of a one-on-one peer mentoring program, either face-to-face or by telephone.
  Interventions: Behavioral: One-on-one peer support
- Control - Standard of care (Active Comparator): "Standard of care" is at the discretion of the treating rheumatologist.
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: One-on-one peer support — The peer support intervention will take the form of a one-on-one peer mentoring program, using a mutually agreed upon method of communication between each pair of peer mentor and EIA participant (either by telephone or face-to-face meeting at a neutral public location). The research team will pair trained peer mentors and individuals with EIA as closely as possible based on such characteristics as sex, age, working status, and specific disease/type of IA. Peer mentors will be responsible to initiate and maintain contact with individuals with EIA. Individuals with EIA and peer mentors will be asked to have contact once a week for 30 minutes during the 12-week study period. Meetings/ interactions will not be prescribed; rather they will be defined by the individual with EIA. Peer mentors will provide support based on the needs of the individual they are mentoring. As such the nature of each interaction is likely to vary among pairs and from one interaction to the next.
  Arms: One-on-one peer support
Behavioral: Standard of care — "Standard of care" is at the discretion of the treating rheumatologist. In addition to information and patient education about the underlying disease process provided at the time of diagnosis, it may include referral to allied health professionals (e.g., physiotherapist, occupational therapist, podiatrist, social worker). This may be via referral to The Arthritis Society or directly to individual practitioners. In addition, it may include referral to voluntary support programs in the community (e.g., Arthritis Self-Management Program).
  Arms: Control - Standard of care

SUMMARY:
Peer support (including informational, emotional, appraisal support) has been shown to help persons with chronic conditions. The goal of this research is to examine the impact of early peer support on the health and quality of life of individuals with early inflammatory arthritis (EIA). The investigators hypothesize that early peer support will result in improved use of disease modifying anti-rheumatic drug (DMARD) or biologic treatment, self-efficacy, coping efficacy, social support, health-related quality of life, self-management, and disease activity score as well as reduced anxiety for individuals with EIA within two years of their diagnosis. In this study, persons with IA will be trained as peer mentors using a training program developed for a pilot study. Individuals with EIA will be randomized to receive either "peer support program" or "standard care". Peer mentors will be paired with a person with EIA to provide one-on-one support (face-to-face or telephone) once a week for approximately 30 minutes over a 12-week period. All "standard care" participants will receive the peer mentoring intervention at the end of study. Both groups will be evaluated using self-administered questionnaires and clinical assessments, and results of the two groups will be compared. This information will be used to design a larger study.

DETAILED DESCRIPTION:
Background: The investigators are proposing to examine the effectiveness of a peer support program, the aim of which is to assist individuals with early inflammatory arthritis (EIA) to receive the education and support they need to make decisions to manage their disease. Peer support (including informational, emotional, appraisal support) has been shown to assist persons with chronic conditions and may address challenges with receiving timely and proper treatment in persons with EIA.

Purpose: The goal of this pilot randomized controlled trial (RCT) is to evaluate the effectiveness of peer support to improve the health and quality of life of individuals with EIA. The investigators hypothesize that early peer support will result in improved use of treatment, self-efficacy, coping efficacy, social support, health-related quality of life, self-management, and disease activity score, as well as reduced anxiety for individuals with EIA within two years of their diagnosis.

Methods: This proposal builds on a pilot study, currently underway, to develop and evaluate the acceptability and feasibility of a peer support intervention for persons with EIA. The proposed effectiveness study will employ a RCT design with a wait list control group. Individuals with IA (diagnosis 2 or more years) will be trained as peer mentors using the revised pilot study training program. Peer mentors will be matched with a person newly diagnosed with IA to provide one-on-one support (face-to-face or telephone) over a 12-week period. Individuals with EIA will be recruited from rheumatology clinics at Sunnybrook Health Sciences Centre and Mount Sinai Hospital. Individuals with EIA will be randomized to either "intervention" or "standard care" (wait list). All "standard care" participants with EIA will receive the peer mentoring program at the end of study period; their outcomes will be also be evaluated. Both "intervention" and "standard care" participants will complete clinical assessments and self-administered questionnaires before and after (immediate post-program and 3-month follow-up) study completion to evaluate use of treatment, self-efficacy, coping efficacy, social support, health-related quality of life, anxiety, self-management, and disease activity count.

Implication: The study aims to improve the education and support for patients with EIA. The data from this study will be used to further refine the intervention and study design to be subsequently submitted for further effectiveness testing in a larger scale RCT.

ELIGIBILITY:
Inclusion Criteria:

* EIA disease (rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis) duration 6 - 52 weeks
* At least 3 swollen joints, assessed by the treating rheumatologist, OR Positive compression test for the metacarpophalangeal joints, OR Positive compression test for the metatarsophalangeal joints, OR At least 30 minutes of morning stiffness (Lineker et al., 1999)
* Prescription of a DMARD/biologic by the treating rheumatologist
* Ability to speak, understand, read and write English without the aid of a secondary support person
* Ability to provide informed consent

Exclusion Criteria:

• Diagnosis of osteoarthritis, Systemic lupus erythematosus, DM neuropathy or trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-05 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Use of orally administered DMARD or biologic treatment | 0 months (baseline), immediate post-program, 3 months post-program
  Use of orally administered DMARD or biologic treatment in individuals with EIA as determined indirectly through the modified Morisky scale for medication adherence

SECONDARY OUTCOMES:
Self-efficacy | 0 months (baseline), immediate post-program, 3 months post-program
  Self-efficacy using Self-Efficacy for Managing Chronic Disease 6-Item Scale (SES)
Health-related quality of life | 0 months (baseline), immediate post-program, 3 months post-program
  Health-related quality of life as measured by the Arthritis Impact Measurement Scales, 2nd edition (AIMS2
Anxiety | 0 months (baseline), immediate post-program, 3 months post-program
  Anxiety is measured by the Arthritis Impact Measurement Scales, 2nd edition (AIMS2), dimension sub score for anxiety
Coping-efficacy | 0 months (baseline), immediate post-program, 3 months post-program
  Coping-efficacy as assessed using a measure developed by Gignac et al. (2000)
Social support | 0 months (baseline), immediate post-program, 3 months post-program
  Social support as measured by Medical Outcomes Study Social Support Survey (MOSSS)
Self-management | 0 months (baseline), immediate post-program, 3 months post-program
  Self-management as evaluated using Patient Activation Measure (PAM) to measure the knowledge, skills, and confidence aspects of self management
Disease activity | 0 months (baseline), immediate post-program, 3 months post-program
  Disease activity as assessed using the Clinical Disease Activity Index (CDAI): A rheumatologist from the research team will conduct clinical assessments for CDAI score, which is a propensity score for disease activity in rheumatoid arthritis. It accounts for upper extremity tender and swollen joints, and patient and evaluator impressions of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Bell, MD, FRCPC, Principal Investigator — Division of Reumatology, Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario